CLINICAL TRIAL: NCT02916901
Title: A Randomized, Double-blind, Placebo-controlled, Multiple Dosing, Cross-over Phase I Clinical Trial to Investigate the Effect of CKD-519 on 24-h Ambulatory Blood Pressure After Oral Administration in Healthy Adult Volunteers
Brief Title: Study to Investigate the Influence of CKD-519 on 24-h Ambulatory Blood Pressure in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 148HPS16006
Record Dates: First submitted 2016-09-20; First posted 2016-09-28 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2016-09

CONDITIONS: Healthy Volunteers
Keywords: Dyslipidemia; CKD-519; CETP inhibitor; ABPM
MeSH Terms: conditions — Dyslipidemias | interventions — CKD-519

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CKD-519 200mg (Experimental): CKD-519 tab(formulation II) 200mg (100mg X 2tabs)
  Interventions: Drug: CKD-519 200mg
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CKD-519 200mg
  Other Names: (formulation II) 200mg (100mg X 2tabs)
  Arms: CKD-519 200mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine influence of CKD-519 on 24-h ambulatory blood pressure after oral administration in healthy adult volunteers.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled, multiple dosing, cross-over phase I clinical trial to investigate the effect of CKD-519 on 24-h ambulatory blood pressure after oral administration in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Between 19 aged and 55 aged in healthy adult
2. Body weight more than 55kg in male, 50kg in female
3. Body Mass Index more than 18.5 and under 25(body mass index=kg/m2)
4. If female, must include more than one among the items

   * The menopause(there is no natural menses for at least 2 years)
   * Surgical Infertility(hysterectomy or bilateral oophorectomy, tubal ligation or other methods of infertility condition
5. If men has sexual life with women of childbearing age, Necessarily he agrees that use condoms and do not sperm donation until two months during clinical trials and after the final dosage of investigational products
6. Those who fully understand about this clinical trials after enough hearing, and then decided to join the clinical trials by themselves and to comply with the precautions written consent.

Exclusion Criteria:

1. Have clinically significant disease that hepatobiliary system(severe hepatic impairment, etc), kidney(severe renal impairment, etc), nervous system, immune system, respiratory system, endocrine system, hemato-oncology disease, cardiovascular system(heart failure, etc) or mental illness, or a history of mental disease.
2. Have a gastrointestinal disease history that can effect drug absorption(Crohn's disease, ulcers, etc.) or surgery(except simple appendectomy or hernia surgery)
3. Hypersensitivity reaction or clinically significant hypersensitivity reaction in the history of drugs or additives.
4. An impossible one who participates in clinical trial including screening tests(medical history taking, BP, 12-lead ECG, physical examination, blood&urine laboratory test result) before 28 days the taking investigational Products.
5. Defined by the following laboratory parameters

   * AST, ALT>1.25 upper limit of normal range
   * Total bilirubin>1.5 upper limit of normal range
   * CPK>1.5 upper limit of normal range
   * eGFR(using by MDRD method)<60mL/min/1.73m2
6. Sitting SBP > 140mmHg or < 90mmHg, sitting DBP > 90mmHg or < 60mmHg, after 5 minutes break.
7. The difference in DBP>10mmHg or SBP >20mmHg at the screening period
8. Drug abuse or have a history of drug abuse shows a positive for urine drug test.
9. Pregnant or lactating women.
10. A heavy caffeine consumer(caffeine>5 cups/day), alcohol consumer(alcohol>210g/week),
11. smoker(except the one who have stopped smoking more than 90days before beginning of study treatment)
12. Subject takes ethical drug or herbal medicine within 14 days, OTC within 7 days before the beginning of study treatment but investigator determine that the taking drug affect this study or could affect the safety of subjects.
13. Subject who takes inhibitor and inducers of drug metabolizing enzyme(Barbiturates etc.) within 30 days.
14. Taking foods containing grapefruit within 7 days before the beginning of study treatment(ex. Drinking containing grapefruit of 1L per a day or more within 7 days before the beginning of study treatment)
15. Subject who treated with any investigational drugs within 90 days before the beginning of study treatment
16. Previously donate whole blood within 60 days or component blood within 30 days.
17. Positive for Serology test(Hepatitis B, Hepatitis C, HIV)
18. An impossible one who participants in clinical trial by investigator's decision including laboratory test result or another reason

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change in 24h average SBP and DBP from baseline to Day 14 Each time point is as following: Daytime: 06:00~21:59 Nighttime: 22:00~05:59 | 14days

SECONDARY OUTCOMES:
Cmax,ss of CKD-519 | 0(predose)~24 at day15
AUCτ,ss of CKD-519 | 0(predose)~24 at day15
Tmax,ss of CKD-519 | 0(predose)~24 at day15

CONTACTS AND LOCATIONS:
Overall Officials: Min Soo Park, MD, PhD, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, Seodaemun-gu 120-752, South Korea

IPD SHARING:
Plan to Share IPD: No